CLINICAL TRIAL: NCT01177644
Title: Safety and Preliminary Efficacy Study of PDS-1.0 in Patients With Neovascular AMD
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Forsight Vision4 (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FSV4 FH-1
Record Dates: First submitted 2010-08-05; First posted 2010-08-09 (Estimated); Last update posted 2012-08-22 (Estimated); Status verified 2012-08

CONDITIONS: Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

ARMS (1):
- Active (Experimental)
  Interventions: Drug: PDS 1.0

INTERVENTIONS:
Drug: PDS 1.0

SUMMARY:
This study will evaluate the safety and preliminary effectiveness of PDS 1.0 in patients with neovascular AMD.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of CNV secondary to AMD confirmed by fluorescein angiography, not previously treated
* Retinal thickness due to edema of at least 300um in the study eye
* Best corrected visual acuity of 20/80 or worse in the study eye
* Best corrected visual acuity of 20/40 or better in the fellow eye

Exclusion Criteria:

* Evidence of scarring CNV (e.g. geographic atrophy) in the study eye
* Fibrosis >75% of lesion area in the study eye

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-01; Primary Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
Change in retinal thickness measured by Optical Coherence Tomography | Monthly

SECONDARY OUTCOMES:
Change in Best Corrected Visual Acuity | Monthly

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv, Israel